CLINICAL TRIAL: NCT02801630
Title: An Evaluation of the Effect of a Surface Acoustic Wave Patch Device on the Symptons of Trigeminal Neuralgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rosenblum, Jonathan I., DPM (Individual)
Collaborators: Nanovibronix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USTN1
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Crossover (Sham Comparator): After the enrollment and lead in period, subjects will be given a sham device to sleep with every night for a month. They will be asked to fill out their pain and analgesic use logs, and undergo the bi weekly assessments. After a month they will be crossed over to an active "Painshield SAW patch device" and will continue to complete their pain and analgesic use logs as well as undergo biweekly assessments for months two and 3.
  Interventions: Device: PainShield SAW Patch Device
- Active Device (Active Comparator): After the enrollent and lead in period, subjects will be given an active PainSHield SAW Patch device to sleep with every night. They will be asked to fill out their pain and analgesic use logs, and undergo bi weekly assessments. They will continue to use the device while completing their logs and undergoing assessments for 3 months.
  Interventions: Device: PainShield SAW Patch Device

INTERVENTIONS:
Device: PainShield SAW Patch Device — The PainShield is a self contained Surface Acoustic Wave device, where the waves are delivered locally through a trasnducer embedded into a patch that sits on the affected area.

SUMMARY:
This is a double blinded randomized control trial of a Surface Acoustic Wave Patch device for the treatment of Trigeminal Neuralgia. This will be a crossover study for the group that receives the sham device. Subjects will be monitored for subjective criteria of pain and quality of life, as well as objective measurement of analgesic usage.

DETAILED DESCRIPTION:
This study is a double blinded randomized control trial of a Surface acoustic wave patch device for the treatment of Trigeminal Neuralgia. All subjects will be enrolled for a 14 day lead up period, where baseline measures of pain, quality of life and analgesic use will be recorded.

During the first month of the study subjects will be randomized into a sham or active device group. Both groups will be assessed every two weeks for pain, quality of life and analgesic use. After 4 weeks, those subjects in the sham group will be crossed over into the active group. Both groups will continue to be assessed biweekly through months 2 and 3.

After 3 months of treatment a final assessment will be conducted and the results evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with trigeminal neuralgia refractory to medical treatment (modified BNI V).

Exclusion Criteria:

* Male or female, under the age of 18. Active illicit drug use Pregnancy. Psychiatric illness which may prevent the patient from participation in the study.

Anesthesia dolorosa with pain greater than or equal to 3/10 Dental implants. Other known pathology of the trigeminal nerve including iatrogenic anesthesia dolorosa.

Cancer and bone metastases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pain | 90 days
  The Patients level of pain will be assessed by Visual Analog Scale daily

SECONDARY OUTCOMES:
Quality of Life | 90 days
  The patients satisfaction and quality of life will be measured by questionnaires including the SF-36
Rescue Drug Use | 90 days
  The patients use of rescue medication will be recorded during the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: William Stern, Study Director — Sponsor Representative
Locations (1):
- NanoVibronix, Elmsford, New York, United States

IPD SHARING:
Plan to Share IPD: No